CLINICAL TRIAL: NCT00972244
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase 2 Trial to Evaluate the Efficacy and Safety of Dapagliflozin as Monotherapy in Japanese Subjects With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control
Brief Title: Trial to Evaluate the Efficacy and Safety of Dapagliflozin in Japanese Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D1692C00005
Record Dates: First submitted 2009-08-31; First posted 2009-09-04 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Japanese; phase 2; efficacy; safety; dapagliflozin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): 1mg dapagliflozin
  Interventions: Drug: Dapagliflozin
- 2 (Experimental): 2.5mg dapagliflozin
  Interventions: Drug: Dapagliflozin
- 3 (Experimental): 5mg dapagliflozin
  Interventions: Drug: Dapagliflozin
- 4 (Experimental): 10mg dapagliflozin
  Interventions: Drug: Dapagliflozin
- 5 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — once daily, 12 weeks
  Arms: 1; 2; 3; 4
Drug: Placebo — once daily, 12 weeks
  Arms: 5

SUMMARY:
The purpose of this study is to obtain information on efficacy and safety of dapagliflozin in Japanese patients with Type 2 Diabetes. This will be done by comparing the effect of dapagliflozin to placebo when given in oral doses.

ELIGIBILITY:
Inclusion Criteria:

* Japanese Subjects with type 2 diabetes mellitus.
* Strictly/relatively treatment naïve Subjects with HbA1c ≥ 7.0% and ≤ 10%, or Subjects treated with single or two (less than half of the approved maximal dose for each) oral anti-hyperglycaemic agent with HbA1c ≤ 8%.
* Provision of informed consent.

Exclusion Criteria:

* Having clinically relevant medical history or concurrent disease such as cardiovascular disease, renal disease, retinopathy, hepatic disease and haematological disease.
* The investigator(s) judged that the Subject should not participate in the study according to screening test or medical history.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parikh Shamik, Study Director — AstraZeneca
Locations (20):
- Japan (20):
  - Research Site, Anjyo
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Daitō
  - Research Site, Kamagaya
  - Research Site, Kashiwara
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Naka
  - Research Site, Nakano
  - Research Site, Nerima-ku
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Shibuya-ku
  - Research Site, Shinjyuku-ku
  - Research Site, Suita
  - Research Site, Uji
  - Research Site, Wakayama
  - Research Site, Yamato

REFERENCES:
- [Derived] Kohan DE, Fioretto P, Johnsson K, Parikh S, Ptaszynska A, Ying L. The effect of dapagliflozin on renal function in patients with type 2 diabetes. J Nephrol. 2016 Jun;29(3):391-400. doi: 10.1007/s40620-016-0261-1. Epub 2016 Feb 19. PMID 26894924

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment: 417; randomized: 279 Study Start Date: August 2009 Study Completion Date: May 2010 Primary Completion Date: May 2010
Groups:
- 1mg Dapagliflozin: Dapagliflozin tablet 1 mg once daily
- 2.5mg Dapagliflozin: Dapagliflozin tablet 2.5 mg once daily
- 5mg Dapagliflozin: Dapagliflozin tablet 5 mg once daily
- 10mg Dapagliflozin: Dapagliflozin tablet 10 mg once daily
- Placebo: Placebo Comparator
Period: Overall Study
Arm/Group | 1mg Dapagliflozin | 2.5mg Dapagliflozin | 5mg Dapagliflozin | 10mg Dapagliflozin | Placebo
Started | 59 | 56 | 58 | 52 | 54
Completed | 54 | 51 | 56 | 52 | 45
Not Completed | 5 | 5 | 2 | 0 | 9
Not completed — Incorrect Enrolment | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0
Not completed — Subject No Longer Meets Study Criteria | 2 | 2 | 0 | 0 | 5
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 0 | 1
Not completed — Safety | 0 | 0 | 0 | 0 | 1
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Various | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set defined as all randomised participants (as randomized) who received at least one dose of double-blind study medication, who have a non-missing baseline value and at least one post-baseline efficacy value for at least one efficacy variable during double-blind period.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1mg Dapagliflozin | 2.5mg Dapagliflozin | 5mg Dapagliflozin | 10mg Dapagliflozin | Placebo | Total
Number analyzed (Participants) | 59 | 56 | 58 | 52 | 54 | 279
Age Continuous [Mean (Standard Deviation); unit: years] | 55.9 (9.73) | 57.7 (9.33) | 58.0 (9.50) | 56.5 (11.47) | 58.4 (9.97) | 57.3 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 11 | 13 | 11 | 64
  Male | 47 | 39 | 47 | 39 | 43 | 215
Race/Ethnicity, Customized [Number; unit: Participants]
  Japanese | 59 | 56 | 58 | 52 | 54 | 279
HBA1C [Mean (Standard Deviation); unit: percent] | 8.10 (0.785) | 7.92 (0.740) | 8.05 (0.660) | 8.18 (0.690) | 8.12 (0.714) | 8.07 (0.720)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change in HbA1c Levels
Description: The primary efficacy endpoint is the absolute change in HbA1c from baseline to Week 12 or the last post-baseline measurement prior to Week 12, if no Week 12 assessment is available.
Time Frame: Baseline to Week 12
Population: Full Analysis Set, participants with non-missing baseline and Week 12 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | 1mg Dapagliflozin | 2.5mg Dapagliflozin | 5mg Dapagliflozin | 10mg Dapagliflozin | Placebo
Number analyzed (Participants) | 59 | 54 | 58 | 52 | 52
percent | -0.12 [-0.25 to 0.01] | -0.10 [-0.24 to 0.04] | -0.37 [-0.50 to -0.23] | -0.44 [-0.58 to -0.29] | 0.35 [0.21 to 0.49]
Statistical Analysis 1: Comparison: 1mg Dapagliflozin vs Placebo; The null hypothesis is given as H0: mean(treat) minus mean(placebo) = 0 versus HA: mean(treat) minus mean(placebo) =/= 0 (with alpha = 0.015 applying Dunnett's adjustment, two-sided); Test type: Superiority or Other; p < 0.0001, ANCOVA — significant at alpha=0.015 (2-sided) applying Dunnett's adjustment. A sequential closed testing procedure was used to control Type I error rate across the primary and key secondary endpoints; with treatment group (all treatment groups included) as fixed effect and baseline value as covariate; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.67 to -0.28], Standard Error of Mean 0.0987
Statistical Analysis 2: Comparison: 2.5mg Dapagliflozin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; with treatment group (all treatment groups included) as fixed effect and baseline value as covariate; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.65 to -0.26], Standard Error of Mean 0.1009
Statistical Analysis 3: Comparison: 5mg Dapagliflozin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; with treatment group (all treatment groups included) as fixed effect and baseline value as covariate; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-0.92 to -0.53], Standard Error of Mean 0.0990
Statistical Analysis 4: Comparison: 10mg Dapagliflozin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; with treatment group (all treatment groups included) as fixed effect and baseline value as covariate; Mean Difference (Final Values) = -0.79, 95% CI 2-sided [-0.99 to -0.59], Standard Error of Mean 0.1018

2. Secondary Outcome: Adjusted Mean Change in Fasting Plasma Glucose
Description: Change in fasting plasma glucose from baseline to Week 12 or the last post-baseline measurement prior to Week 12, if no Week 12 assessment is available.
Time Frame: Baseline to Week 12
Population: Full Analysis Set, participants with non-missing baseline and Week 12 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | 1mg Dapagliflozin | 2.5mg Dapagliflozin | 5mg Dapagliflozin | 10mg Dapagliflozin | Placebo
Number analyzed (Participants) | 50 | 52 | 51 | 47 | 50
mg/dL | -16.63 [-23.25 to -10.00] | -19.97 [-26.47 to -13.47] | -23.49 [-30.06 to -16.93] | -31.92 [-38.76 to -25.09] | 9.45 [2.82 to 16.08]
Statistical Analysis 1: Comparison: 1mg Dapagliflozin vs Placebo; The null hypothesis is given as H0: mean(treat) minus mean(placebo) = 0 versus HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p < 0.0001, ANCOVA — significant at alpha=0.05 (2-sided). Primary and key secondary endpoints are tested following a sequential closed testing procedure within treatment group; with treatment group (all treatment groups included) as fixed effect and baseline value as covariate; Mean Difference (Final Values) = -26.08, 95% CI 2-sided [-35.45 to -16.70], Standard Error of Mean 4.7589
Statistical Analysis 2: Comparison: 2.5mg Dapagliflozin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; with treatment group (all treatment groups included) as fixed effect and baseline value as covariate; Mean Difference (Final Values) = -29.42, 95% CI 2-sided [-38.70 to -20.14], Standard Error of Mean 4.7100
Statistical Analysis 3: Comparison: 5mg Dapagliflozin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; with treatment group (all treatment groups included) as fixed effect and baseline value as covariate; Mean Difference (Final Values) = -32.94, 95% CI 2-sided [-42.28 to -23.60], Standard Error of Mean 4.7402
Statistical Analysis 4: Comparison: 10mg Dapagliflozin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; with treatment group (all treatment groups included) as fixed effect and baseline value as covariate; Mean Difference (Final Values) = -41.37, 95% CI 2-sided [-50.90 to -31.85], Standard Error of Mean 4.8358

3. Secondary Outcome: Proportion of Participants Achieving Glycemic Response Defined as HbA1c <7%
Description: Proportion of participants achieving therapeutic glycemic response defined as glycosylated hemoglobin <7%, after 12 weeks of double-blind therapy
Time Frame: At Week 12
Population: Full Analysis Set, participants with non-missing baseline and week 12 (LOCF) values
Measure: Number; unit: Percentage of participants
Arm/Group | 1mg Dapagliflozin | 2.5mg Dapagliflozin | 5mg Dapagliflozin | 10mg Dapagliflozin | Placebo
Number analyzed (Participants) | 59 | 54 | 58 | 52 | 52
Percentage of participants | 1.7 | 9.3 | 5.2 | 9.6 | 1.9
Statistical Analysis 1: Comparison: 1mg Dapagliflozin vs Placebo; H0: proportion(treat) minus proportion(placebo) = 0 versus HA: proportion(treat) minus proportion(placebo) =/= 0; Test type: Superiority or Other; p = 1.0000, Fisher Exact — not significant at alpha=0.05 (2-sided). Primary and key secondary endpoints are tested following a sequential closed testing procedure within treatment group; Risk Difference (RD) = -0.2, 95% CI 2-sided [-9.1 to 7.6]
Statistical Analysis 2: Comparison: 2.5mg Dapagliflozin vs Placebo; H0: proportion(treat) minus proportion(placebo) = 0 versus HA: proportion(treat) minus proportion(placebo) =/= 0; Test type: Superiority or Other; p = 0.2057, Fisher Exact — [p-value comment as in outcome 3, analysis 1]; Risk Difference (RD) = 7.3, 95% CI 2-sided [-2.3 to 18.8]
Statistical Analysis 3: Comparison: 5mg Dapagliflozin vs Placebo; H0: proportion(treat) minus proportion(placebo) = 0 versus HA: proportion(treat) minus proportion(placebo) =/= 0; Test type: Superiority or Other; p = 0.6203, Fisher Exact — [p-value comment as in outcome 3, analysis 1]; Risk Difference (RD) = 3.2, 95% CI 2-sided [-6.2 to 13.2]
Statistical Analysis 4: Comparison: 10mg Dapagliflozin vs Placebo; H0: proportion(treat) minus proportion(placebo) = 0 versus HA: proportion(treat) minus proportion(placebo) =/= 0; Test type: Superiority or Other; p = 0.2050, Fisher Exact — [p-value comment as in outcome 3, analysis 1]; Risk Difference (RD) = 7.7, 95% CI 2-sided [-2.0 to 19.5]

ADVERSE EVENTS:
Time Frame: Non-serious / serious adverse events on or after the first day and on or prior to the last day of the 12-week double-blind treatment plus 4/30 days or up to the follow-up visit if earlier.
Description: Participants were questioned at each study visit about the occurrence of any health problems and any examination conducted at the study visit was assessed in comparison to the status at study entry.
Arm/Group | 1mg Dapagliflozin | 2.5mg Dapagliflozin | 5mg Dapagliflozin | 10mg Dapagliflozin | Placebo
Serious Adverse Events (participants affected / at risk) | 2/59 | 1/56 | 2/58 | 1/52 | 0/54
Other Adverse Events (participants affected / at risk) | 14/59 | 13/56 | 14/58 | 13/52 | 14/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1mg Dapagliflozin (N=59) | 2.5mg Dapagliflozin (N=56) | 5mg Dapagliflozin (N=58) | 10mg Dapagliflozin (N=52) | Placebo (N=54)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
MULTI-ORGAN FAILURE (General disorders) | 1 | 0 | 0 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
SEPSIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
DERMAL CYST (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1mg Dapagliflozin (N=59) | 2.5mg Dapagliflozin (N=56) | 5mg Dapagliflozin (N=58) | 10mg Dapagliflozin (N=52) | Placebo (N=54)
Constipation (Gastrointestinal disorders) | 3 | 0 | 2 | 0 | 1
Nasopharyngitis (Infections and infestations) | 12 | 10 | 7 | 12 | 13
Headache (Nervous system disorders) | 0 | 3 | 2 | 1 | 0
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3

LIMITATIONS AND CAVEATS:
If an efficacy measurement was unavailable at the time point for analysis, last observation was carried forward (LOCF).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator requests permission to publish data from this study any such publication is to be agreed with AstraZeneca (AZ) in advance. The investigator agrees to provide AZ as soon as possible with drafts of proposed publications. Unless otherwise agreed, AZ shall have a period of 60 days from receipt of the proposed final manuscript to review it and may within such time require that submission for publication of the manuscript be delayed in order for AZ to file patent applications.